CLINICAL TRIAL: NCT05285904
Title: Kesimpta® (Ofatumumab) in Swiss Multiple Sclerosis Patients - an Observational Study (KOSMOS)
Brief Title: Kesimpta® (Ofatumumab) in Swiss Multiple Sclerosis Patients - an Observational Study
Acronym: KOSMOS
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GCH01
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: NIS; Multiple sclerosis; MS; KOSMOS; Ofatumumab; Kesimpta
MeSH Terms: conditions — Multiple Sclerosis | interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ofatumumab: Population under routine medical care prescribed Ofatumumab in an early Relapsing Multiple Sclerosis
  Interventions: Other: Ofatumumab

INTERVENTIONS:
Other: Ofatumumab — Prospective observational cohort study. There is no treatment allocation. Patients administered Ofatumumab, that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This is a multi-center, observational study carried out in Switzerland that aims to describe the effects of Ofatumumab in a setting of routine medical care.

DETAILED DESCRIPTION:
This non-interventional study will observe the effect of Ofatumumab treatment compared to the standard of care (SoC) arm of a closely monitored phase-IIIb study (STHENOS-COMB157G3301) in MS patients in a real-world setting in Switzerland over an observational period of 12 month.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before participating in the study.
2. Diagnosis of RMS per McDonald Criteria (2017) occurred within 3 years prior to initiation of Ofatumumab.
3. Adult patients who have been on treatment with Ofatumumab for at least 3 months, but not longer than 12 months prior to inclusion in the study.
4. Ofatumumab treatment in line with the Swiss Kesimpta® label (i.e. adult patients with active, relapsing forms of MS)
5. Patient is willing and able to complete patient diary during course of the study, as well as to complete PRO questionnaires.

Exclusion Criteria:

1. Use of investigational drugs during the study, OR between Ofatumumab initiation and inclusion into the study, OR within 3 months before Ofatumumab initiation, OR within 5 half-lives of investigational drug before Ofatumumab initiation, OR until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
2. Subjects who are not able to provide consent due to incapable judgement

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include male and female patients (aged ≥ 18 years) with a documented diagnosis of RMS and treated for at least 3 months with Ofatumumab
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with no evidence of disease activity (NEDA-3) | Month 12
  No evidence of disease activity (NEDA-3), as defined by no confirmed MS relapse, no new or enlarging T2 lesions, no Gadolinium-positive T1 lesions, and no six-month confirmed disability worsening, as compared to the SoC arm of STHENOS.

SECONDARY OUTCOMES:
Proportion of patients demonstrating NEDA-3 | Month 12
  Proportion of patients demonstrating NEDA-3 and its components in relation to the Ofatumumab arm of STHENOS.
Proportion of patients demonstrating no evidence of disease activity in individual components of NEDA-3 | Month 12
  Proportion of patients demonstrating no evidence of disease activity in individual components of NEDA-3:
  * No confirmed MS relapse
  * No new or enlarging T2 lesions
  * No Gadolinium-positive T1 lesions
  * No six-month confirmed disability worsening
Proportion of patients with previous DMT medication | Baseline
  Proportion of patients with previous Disease-modifying Therapy (DMT) medication will be collected
Proportion of patients with clinical and MRI parameters | Baseline
  Proportion of patients with Magnet Resonance Imaging (MRI) and clinical parameters will be collected.
  Clinical parameters includes number of T2-hyperintense lesions, T1-contrast-enhancing lesions; number of MS relapse; Extended disability status scale (EDSS)
Proportion of Ofatumumab doses not completed | Month 12
  Proportion of Ofatumumab doses not completed and reason for not completion within 14 days of expected date.
Proportion of participants with a cumulative treatment interruption of more than six months | Month 12
  Proportion of participants with a cumulative treatment interruption of more than six months, calculated as 6 doses not completed.
Adherence to Ofatumumab | Month 12
  Proportion of participants with and without 100% adherence, defined as no dose administered outside of 14 days of expected date
Proportion of patients permanently discontinuing Ofatumumab | Month 12
  Proportion of patients permanently discontinuing Ofatumumab during the study, and reasons for discontinuation.
Interdependency of adherence and clinical outcome in terms of NEDA-3 | Month 12
  Correlation between adherence and clinical outcome in terms of NEDA-3 activity to be measured
Treatment effect of Ofatumumab on the impact of multiple sclerosis as measured by MSIS-29 | Month 12
  The Multiple Sclerosis Impact Scale (MSIS-29) Questionnaire is a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 5 response options. Higher scores reflect greater impact on day to day life
Treatment satisfaction with Ofatumumab as measured by TSQM-9 | Month 12
  The TSQM-9 is a patient questionnaire assessing treatment satisfaction with Ofatumumab.
  It consists of 3 subscales: effectiveness, convenience and global satisfaction. Each scale score was calculated by summing individual items and then transformed to a 0-100 scale. Higher summary scores indicate better satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- Switzerland (12):
  - Novartis Investigative Site, Baden, Canton of Aargau
  - Novartis Investigative Site, Lucerne, Canton of Lucerne
  - Novartis Investigative Site, Sargans, Canton of St. Gallen
  - Novartis Investigative Site, Gland, Canton of Vaud
  - Novartis Investigative Site, Zurich, Canton of Zurich
  - Novartis Investigative Site, Zurich, CHE
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Lucerne
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: No